CLINICAL TRIAL: NCT07307586
Title: A Small Prospective Clinical Study on Azvudine Tablets for Treating Chronic Hepatitis B.
Brief Title: A Small Sample Prospective Clinical Study of Azvudine Tablets to Promote Clinical Cure in Patients With Chronic Hepatitis B
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhigang Ren (Other)
Responsible Party: Sponsor-Investigator, Zhigang Ren, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-KY-0607-002
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B; Azvudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — azvudine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAF Group (Active Comparator): CHB patients with TAF treatment
  Interventions: Drug: TAF
- Azvudine Group (Experimental): CHB patients with Azvudine treatment
  Interventions: Drug: AZVUDINE
- IFN α-2a Group (Active Comparator): CHB patients with IFN α-2a treatment
  Interventions: Drug: IFNα-2a

INTERVENTIONS:
Drug: AZVUDINE — CHB patients with Azvudine treatment
  Arms: Azvudine Group
Drug: TAF — CHB patients with TAF treatment
  Arms: TAF Group
Drug: IFNα-2a — CHB patients with IFNα-2a treatment
  Arms: IFN α-2a Group

SUMMARY:
Through regular monitoring of viral load, liver function and immune cell activity, the long-term efficacy of Adefovir in controlling HBV is precisely evaluated. By employing a dual mechanism of "antiviral action plus immune activation", it offers a novel therapeutic option for achieving clinical cure in chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet the following criteria to be eligible for inclusion in the trial:

  1. Meet the diagnostic criteria for viral hepatitis as outlined in the Chinese Medical Association's Hepatology Branch Guidelines for the Prevention and Treatment of Chronic Hepatitis B, with patients demonstrating sustained positivity for hepatitis B e antigen (HBeAg) and hepatitis B surface antigen (HBsAg) for at least six months;
  2. HBV DNA load > 20,000 copies/mL and HBsAg < 1,500 IU/mL;
  3. Serum alanine aminotransferase (ALT) > 2 times the upper limit of normal;
  4. No prior antiviral therapy prior to hospital admission.

Exclusion Criteria:

* All subjects meeting any of the following criteria shall be excluded from this study:

  1. Individuals co-infected with other hepatotropic viruses, such as hepatitis A, C, D, or E viruses, or HIV;
  2. Patients with concomitant liver metabolic disorders, cirrhosis, autoimmune-related diseases, or other chronic conditions;
  3. Pregnant or breastfeeding women, or those planning pregnancy within one year;
  4. Patients who have received or are currently undergoing antineoplastic therapy;
  5. History of alcohol or substance abuse;
  6. Patients currently taking therapeutic medications or health supplements;
  7. Patients who participated in other clinical trials within 30 days prior to enrolment;
  8. Patients with allergic constitutions or hypersensitivity to any drug or component used in this study;
  9. Patients with gastrointestinal disorders that may impair drug absorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Follow-up at 12 months | 12 month
  Taking the medication orally for 12 months.

SECONDARY OUTCOMES:
Adverse events | Up to 30 days (form the date of confirmed CHB)
  Discontinuation of medication due to adverse events or other reasons

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided